CLINICAL TRIAL: NCT01374802
Title: Effect of Multiple Dosing With 240 mg QD BI 201335 on the Steady-state Pharmacokinetics of 800 mg QD Darunavir Coadministered With 100 mg QD Ritonavir (DRV/r) in Healthy Male and Female Volunteers (an Open-label, Multiple-dose, Single Group, Single Fixed Sequence Phase I Study)
Brief Title: Effect of Multiple Dosing With BI 201335 on the Pharmacokinetics of Darunavir Co-administered With Ritonavir in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1220.49; 2011-000505-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-06-08; First posted 2011-06-16 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir; faldaprevir

ARMS (3):
- BI 201335 (Experimental): capsule for oral administration
  Interventions: Drug: BI 201335
- Darunavir 400 mg (Experimental): tablet for oral administration
  Interventions: Drug: Darunavir
- Ritonavir 100 mg (Experimental): tablet for oral administration
  Interventions: Drug: Ritonavir

INTERVENTIONS:
Drug: Darunavir — 400 mg tablet for oral administration
  Arms: Darunavir 400 mg
Drug: Ritonavir — tablet for oral administration
  Arms: Ritonavir 100 mg
Drug: BI 201335
  Arms: BI 201335

SUMMARY:
The objective of the current study is to investigate the effect of multiple oral daily doses of BI 201335 on the steady-state pharmacokinetics of darunavir co-administered with ritonavir.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects according to the following criteria: medical history, physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age 18 to 55 years (incl.)
3. Body Mass Index (BMI) 18.5 to 29.9 kg/m2 (incl.) and weight greater than 50 kg
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion criteria:

1. Any finding of the medical examination (including blood pressure (BP), pulse rate (PR) and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. History of photosensitivity or recurrent rash.
5. Surgery of the gastrointestinal tract (except appendectomy)
6. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
7. History of relevant orthostatic hypotension, fainting spells or blackouts.
8. Chronic or relevant acute infections
9. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
10. Intake of drugs with a long half-life (more than 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (more than 10 cigarettes)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 30 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. ALT outside the normal range or any other laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of trial site
19. The subject is not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
20. Positive serology tests for Human immunodeficiency virus (HIV) and hepatitis B / C virus
21. Vulnerable subjects (e.g. persons kept in detention)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.49.1 Boehringer Ingelheim Investigational Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: The study was performed as an open-label, multiple-dose, single-group, fixed-sequence study in 14 healthy volunteers.
  Period 1: Darunavir 800 mg once daily coadministered with ritonavir 100 mg (DRV/r).
  Period 2: Faldaprevir together with DRV/r.
Period: Overall Study
Arm/Group | All Subjects
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was performed as an open-label, multiple-dose, single-group, fixed-sequence study in 14 healthy volunteers.
Arm/Group | All Subjects
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: AUCτ,ss of Darunavir
Description: area under the concentration-time curve of the analyte in plasma at steadystate over a uniform dosing interval τ of darunavir.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00,12:00 hours (h) after drug administration on day 8 (DRV/r) and day 16 (BI 201335+DRV/r)
Population: Pharmacokinetic (PK) set: all subjects in the treated set who provided at least one observation for at least one primary endpoint without any important protocol violations relevant to the pharmacokinetic evaluation and who did not experience vomiting at or before 2 times median tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Darunavir+Ritonavir: oral administration of darunavir 800 mg once daily coadministered with ritonavir 100 mg (DRV/r) once daily
- Faldaprevir+Darunavir+Ritonavir: oral administration of Faldaprevir 240 mg once daily together with DRV/r. Faldaprevir 480 mg loading dose together with DRV/r on the first day.
Arm/Group | Darunavir+Ritonavir | Faldaprevir+Darunavir+Ritonavir
Number analyzed (Participants) | 14 | 14
ng*h/mL | 57200 (29.5) | 66000 (39.9)
Statistical Analysis 1: Comparison: Darunavir+Ritonavir vs Faldaprevir+Darunavir+Ritonavir; relative bioavailability comparison (Faldaprevir+DRV/r : DRV/r) of Darunavir; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 115.29, 90% CI 2-sided [101.36 to 131.13], Standard Deviation 19.4 — the standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Cτ,ss of Darunavir
Description: concentration of the analyte in plasma at steady-state after a uniform dosing interval τ=24h of darunavir
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00,12:00 h after drug administration on day 8 (DRV/r) and day 16 (BI 201335+DRV/r)
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Darunavir+Ritonavir | Faldaprevir+Darunavir+Ritonavir
Number analyzed (Participants) | 14 | 14
ng/mL | 1330 (49.5) | 1170 (90.3)
Statistical Analysis 1: Comparison: Darunavir+Ritonavir vs Faldaprevir+Darunavir+Ritonavir; relative bioavailability comparison (Faldaprevir+DRV/r : DRV/r) of Darunavir; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 87.91, 90% CI 2-sided [68.609 to 112.630], Standard Deviation 38.3 — the standard deviation is actually the geometric coefficient of variation

3. Primary Outcome: Cmax,ss of Darunavir
Description: maximum measured concentration of the analyte in plasma at steady-state
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Darunavir+Ritonavir | Faldaprevir+Darunavir+Ritonavir
Number analyzed (Participants) | 14 | 14
ng/mL | 4930 (23.9) | 6330 (26.5)
Statistical Analysis 1: Comparison: Darunavir+Ritonavir vs Faldaprevir+Darunavir+Ritonavir; relative bioavailability comparison (Faldaprevir+DRV/r : DRV/r) of Darunavir; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 128.41, 90% CI 2-sided [115.724 to 142.489], Standard Deviation 15.6 — the standard deviation is actually the geometric coefficient of variation

4. Secondary Outcome: Tmax,ss of Darunavir
Description: time from last dosing to maximum concentration of the analyte in plasma at steady state
Time Frame: as for outcome 1
Population: PK set
Measure: Median (Full Range); unit: h
Arm/Group | Darunavir+Ritonavir | Faldaprevir+Darunavir+Ritonavir
Number analyzed (Participants) | 14 | 14
h | 1.50 (33.9) [1.00 to 3.00] | 2.01 (37.3) [1.00 to 4.00]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) occurring up to 9 days after first drug administration of DRV/r were assigned to the treatment DRV/r and AEs occurring up to 13 days after last drug administration of DRV/r+FDV were assigned to the combined treatment DRV/r+FDV.
Description: The subjects were required to spontaneously report any AEs. In addition, subjects were assessed regularly for AEs during the trial.
Groups:
- Darunavir+Ritonavir: oral administration of darunavir 800 mg once daily coadministered with ritonavir 100 mg (DRV/r)once daily
Arm/Group | Darunavir+Ritonavir | Faldaprevir+Darunavir+Ritonavir
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 7/14 | 11/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darunavir+Ritonavir (N=14) | Faldaprevir+Darunavir+Ritonavir (N=14)
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Fatigue (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.